CLINICAL TRIAL: NCT05110066
Title: Balloon Pulmonary anGiOplasty Versus Pulmonary Endarterectomy in Patients With Chronic ThromboEmbolic Pulmonary Hypertension: a Non-inferiority Randomized Trial
Brief Title: BPA vs. PEA in CTEPH
Acronym: GO-CTEPH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Kerckhoff Klinik (Other); Medical University of Vienna (Other); Papworth Hospital NHS Foundation Trust (Other Government); St. Antonius Hospital (Other); Utrecht University (Other); KU Leuven (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 190580-0002
Record Dates: First submitted 2021-10-04; First posted 2021-11-05 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPA group (Active Comparator): Balloon pulmonary angioplasty. Typically 4-8 sessions are needed to treat the patient. The specific pre-planning protocol, choice of wires and balloons, the number of vessels treated per session, and the decision that no further BPA sessions are needed is at the discretion of the treating physician.
  Interventions: Procedure: Balloon pulmonary angioplasty
- PEA group (Active Comparator): Patients randomized to PEA will undergo surgery within 4 months after randomization and optional run-in phase. Distality of the dissection plane is at the discretion of the operating physicians.
  Interventions: Procedure: Pulmonary endarterectomy

INTERVENTIONS:
Procedure: Pulmonary endarterectomy — Surgical pulmonary endarterectomy is done by a thoracic surgical procedure by removing chronic thrombotic material by intimal dissection with patient on cardiopulmonary bypass.
  Arms: PEA group
Procedure: Balloon pulmonary angioplasty — Percutaneous balloon pulmonary angioplasty is performed using standard percutaneous technique to break the fibrotic clots in the pulmonary arteries using percutaneous transluminal angioplasty balloons.
  Arms: BPA group

SUMMARY:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a rare and potentially life-threatening progressive disease that evolves from unresolved pulmonary embolism. Gold standard treatment for CTEPH is pulmonary endarterectomy (PEA) performed by skilled cardio-thoracic surgeons.

Some patients may not be surgical candidates due to co-morbidities or because the vascular lesions are too distal making them technically inoperable. In these patients, balloon pulmonary angioplasty (BPA) has emerged as an effective treatment. In a subgroup of patients, the distribution of vascular lesions makes it possible to perform either BPA or PEA. There has never been a head-to head comparison of BPA with PEA. The aim of this study is therefore, to evaluate if BPA is non-inferior to PEA in patients with (CTEPH) who are eligible for both treatments.

DETAILED DESCRIPTION:
An investigator-initiated multicenter, prospective, randomized, controlled, open label, non-inferiority trial. The study will randomize (1:1) 152 patients with CTEPH who are eligible for both PEA and BPA. Patients will be screened for study inclusion at the local CTEPH multidisciplinary team conference and eligibility for both PEA and BPA will be confirmed by a central adjudication committee.

PEA or BPA will be completed within 6 months from randomization. Follow-up visit with right heart catheterization will be completed at 4 months and 12 months after PEA or last BPA session.

Primary end-point is change in pulmonary vascular resistance from baseline to 4 months and 12 months after PEA or the last BPA session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic thromboembolic pulmonary hypertension according to current European society of cardiology/European Respiratory Society guidelines and eligible for both pulmonary endarterectomy and ballon pulmonary angioplasty by decision at the local multidisciplinary team conference and central adjudication committee
* Written informed consent from the patient
* Patient age >17 and <80 years
* Able to understand and follow instructions and to participate in the entire study period

Exclusion Criteria:

* Life expectancy <12 months
* Co morbidities evaluated at the multidisciplinary team conference, that contributes significantly to the patients pulmonary hypertension
* Not possible to perform balloon pulmonary angioplasty or pulmonary endarterectomy within 4 months after randomization.
* Evaluated at multidisciplinary team conference that changes in pulmonary artery hypertension targeted therapy between baseline and 4 months follow-up is inevitable*
* Known pregnancy or positive urine Human chorionic gonadotropin screening test in fertile women
* Previous balloon pulmonary angioplasty or pulmonary endarterectomy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance | 4 months and 12 months
  Change in pulmonary vascular resistance from baseline to 4-months and 12-months after the procedure(s). Patients on medical treatments at baseline will remain on medical treatments until the assessment of the primary endpoint, and be taken off if hemodynamics permit

SECONDARY OUTCOMES:
Mean pulmonary artery pressure | 4 months and 12 months
  Mean pulmonary artery pressure measured by right heart catheterization
Cardiac index | 4 months and 12 months
  Cardiac index measured by right heart catheterization
Mean right atrial pressure | 4 months and 12 months
  Right atrial pressure measured by right heart catheterization
Six minutes walking distance | 4 months and 12 months
  Six minutes walking distance
Time to clinical worsening | 4 months and 12 months
  Clinical worsening includes all-cause mortality, nonelective hospitalization for pulmonary artery hypertension, and disease progression (disease progression is defined as a reduction from baseline in the six minutes walking distance by 15% plus worsening functional class (except for patients already in Orld health organization functional class IV).)
N-terminal pro B-type natriuretic peptide | 4 months and 12 months
  N-terminal pro B-type natriuretic peptide
Quality of life evaluated by the "Living with pulmonary hypertension questionnaire" | 4 months and 12 months
  Measured by the use of Living with pulmonary hypertension questionnaire (21 questions scored 0-5. Minimum score is 0 and maximum score is 105. Low score means high quality of life and a high score means a low quality of life).

OTHER OUTCOMES:
Peri-operative/peri-interventional complications | 30 days
  Complications related to balloon pulmonary angioplasty and pulmonary endarterectomy will be recorded
Total length of hospital stay in both groups | 4 month
  Time of hospital stay will be recorded
Median survival at 12 month | 12 months
  Deaths will be recorded recorded and a median 12 month survival will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lang, MD,Prof, Study Chair — Medical University of Vienna; Harm Jan Bogaard, MD, Prof., Study Chair — Amsterdam University Medical Center; Marion Delcroix, MD, Prof., Study Chair — KU Leuven; Marco Post, MD, Prof., Study Chair — St. Antonius Hospital; Gregely Meszaros, MD, Study Chair — Pulmonary Hypertension Association Europe; Johanna Pepke-Zaba, MD, Prof., Study Chair — Papworth Hospital NHS Foundation Trust; Christoph Wiedenroth, MD, Study Chair — Kerckhoff Klinik
Locations (2):
- Aarhus University Hospital, Aarhus, Denmark
- Royal Ppworth, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Lang IM, Pesavento R, Bonderman D, Yuan JX. Risk factors and basic mechanisms of chronic thromboembolic pulmonary hypertension: a current understanding. Eur Respir J. 2013 Feb;41(2):462-8. doi: 10.1183/09031936.00049312. Epub 2012 Jun 14. PMID 22700839
- [Background] Gall H, Hoeper MM, Richter MJ, Cacheris W, Hinzmann B, Mayer E. An epidemiological analysis of the burden of chronic thromboembolic pulmonary hypertension in the USA, Europe and Japan. Eur Respir Rev. 2017 Mar 29;26(143):160121. doi: 10.1183/16000617.0121-2016. Print 2017 Mar 31. PMID 28356407
- [Background] Gerges C, Gerges M, Friewald R, Fesler P, Dorfmuller P, Sharma S, Karlocai K, Skoro-Sajer N, Jakowitsch J, Moser B, Taghavi S, Klepetko W, Lang IM. Microvascular Disease in Chronic Thromboembolic Pulmonary Hypertension: Hemodynamic Phenotyping and Histomorphometric Assessment. Circulation. 2020 Feb 4;141(5):376-386. doi: 10.1161/CIRCULATIONAHA.119.041515. Epub 2020 Jan 3. PMID 31896275
- [Background] Delcroix M, Vonk Noordegraaf A, Fadel E, Lang I, Simonneau G, Naeije R. Vascular and right ventricular remodelling in chronic thromboembolic pulmonary hypertension. Eur Respir J. 2013 Jan;41(1):224-32. doi: 10.1183/09031936.00047712. Epub 2012 Aug 16. PMID 22903956
- [Background] Riedel M, Stanek V, Widimsky J, Prerovsky I. Longterm follow-up of patients with pulmonary thromboembolism. Late prognosis and evolution of hemodynamic and respiratory data. Chest. 1982 Feb;81(2):151-8. doi: 10.1378/chest.81.2.151. PMID 7056079
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Jenkins D, Madani M, Fadel E, D'Armini AM, Mayer E. Pulmonary endarterectomy in the management of chronic thromboembolic pulmonary hypertension. Eur Respir Rev. 2017 Mar 15;26(143):160111. doi: 10.1183/16000617.0111-2016. Print 2017 Jan. PMID 28298388
- [Background] Pepke-Zaba J, Delcroix M, Lang I, Mayer E, Jansa P, Ambroz D, Treacy C, D'Armini AM, Morsolini M, Snijder R, Bresser P, Torbicki A, Kristensen B, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Hamid AM, Jais X, Simonneau G. Chronic thromboembolic pulmonary hypertension (CTEPH): results from an international prospective registry. Circulation. 2011 Nov 1;124(18):1973-81. doi: 10.1161/CIRCULATIONAHA.110.015008. Epub 2011 Oct 3. PMID 21969018
- [Background] Lang I, Meyer BC, Ogo T, Matsubara H, Kurzyna M, Ghofrani HA, Mayer E, Brenot P. Balloon pulmonary angioplasty in chronic thromboembolic pulmonary hypertension. Eur Respir Rev. 2017 Mar 29;26(143):160119. doi: 10.1183/16000617.0119-2016. Print 2017 Mar 31. PMID 28356406
- [Background] Delcroix M, Lang I, Pepke-Zaba J, Jansa P, D'Armini AM, Snijder R, Bresser P, Torbicki A, Mellemkjaer S, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Jais X, Ambroz D, Treacy C, Morsolini M, Jenkins D, Lindner J, Dartevelle P, Mayer E, Simonneau G. Long-Term Outcome of Patients With Chronic Thromboembolic Pulmonary Hypertension: Results From an International Prospective Registry. Circulation. 2016 Mar 1;133(9):859-71. doi: 10.1161/CIRCULATIONAHA.115.016522. Epub 2016 Jan 29. PMID 26826181
- [Background] Khan MS, Amin E, Memon MM, Yamani N, Siddiqi TJ, Khan SU, Murad MH, Mookadam F, Figueredo VM, Doukky R, Benza RL, Krasuski RA. Meta-analysis of use of balloon pulmonary angioplasty in patients with inoperable chronic thromboembolic pulmonary hypertension. Int J Cardiol. 2019 Sep 15;291:134-139. doi: 10.1016/j.ijcard.2019.02.051. Epub 2019 Feb 23. PMID 30850238
- [Background] Tanabe N, Kawakami T, Satoh T, Matsubara H, Nakanishi N, Ogino H, Tamura Y, Tsujino I, Ogawa A, Sakao S, Nishizaki M, Ishida K, Ichimura Y, Yoshida M, Tatsumi K. Balloon pulmonary angioplasty for chronic thromboembolic pulmonary hypertension: A systematic review. Respir Investig. 2018 Jul;56(4):332-341. doi: 10.1016/j.resinv.2018.03.004. Epub 2018 Jul 3. PMID 30008295
- [Background] Kim NH, Delcroix M, Jenkins DP, Channick R, Dartevelle P, Jansa P, Lang I, Madani MM, Ogino H, Pengo V, Mayer E. Chronic thromboembolic pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D92-9. doi: 10.1016/j.jacc.2013.10.024. PMID 24355646
- [Background] Mayer E, Jenkins D, Lindner J, D'Armini A, Kloek J, Meyns B, Ilkjaer LB, Klepetko W, Delcroix M, Lang I, Pepke-Zaba J, Simonneau G, Dartevelle P. Surgical management and outcome of patients with chronic thromboembolic pulmonary hypertension: results from an international prospective registry. J Thorac Cardiovasc Surg. 2011 Mar;141(3):702-10. doi: 10.1016/j.jtcvs.2010.11.024. PMID 21335128